CLINICAL TRIAL: NCT05102396
Title: Topical Oxybutynin Deodorant for Axillary Hyperhidrosis: Local or Systemic Effect? The TODAY Trial
Brief Title: Topical Oxybutynin for Treatment of Hyperidrosis: Local or Systemic Effect?
Acronym: TODAY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samantha Rodrigues Camargo Neves de Moura (Other)
Collaborators: Science Valley Research Institute (Other)
Responsible Party: Sponsor-Investigator, Samantha Rodrigues Camargo Neves de Moura, Samantha Rodrigues Camargo Neves de Moura - Santa Casa de Sao Paulo School of Medical Sciences, Science Valley Research Institute
Organization: Science Valley Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TODAY Trial
Record Dates: First submitted 2021-10-14; First posted 2021-11-01 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Hyperhidrosis; Oxybutynin; Sweat Gland Diseases; Skin Diseases; Autonomic Agents; Cholinergic Antagonists; Parasympatholytics
Keywords: hyperhidrosis; oxybutynin; anticholinergic; axillary hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis; Sweat Gland Diseases; Skin Diseases | interventions — oxybutynin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Topical oxybutynin spray (Experimental): Participants with axillary hyperhidrosis will receive topical oxybutynin spray (10%) in an appropriate dose of 2 puffs in each armpit twice a day for 35 days.
  Interventions: Drug: Topical oxybutynin spray
- Topical placebo spray (Placebo Comparator): Participants with axillary hyperhidrosis will receive topical placebo spray in an appropriate dose of 2 puffs in each armpit twice a day for 35 days.
  Interventions: Drug: Topical placebo spray
- Oral oxybutynin (Active Comparator): Participants with axillary hyperhidrosis will receive oral oxybutynin for 35 days as follows: during the first week, participants will receive 2.5 mg of oxybutynin once a day in the evening; from the 8th to the 14th day, they will receive 2.5 mg twice a day; and from the 15th day to the end of the 35th day of treatment, they will receive 5 mg twice a day.
  Interventions: Drug: Oral oxybutynin

INTERVENTIONS:
Drug: Topical oxybutynin spray — Participants will receive topical oxybutynin spray (10%).
  Arms: Topical oxybutynin spray
Drug: Topical placebo spray — Participants will receive topical placebo spray.
  Arms: Topical placebo spray
Drug: Oral oxybutynin — Participants will receive oxybutynin (tablets).
  Arms: Oral oxybutynin

SUMMARY:
The TODAY trial is a study to evaluate the efficacy and safety of topical oxybutynin deodorant for use in patients with axillary hyperhidrosis.

DETAILED DESCRIPTION:
Background: Anticholinergics, both orally and topically, have been shown to enhance quality of life and reduce sweat in patients with hyperhidrosis, potentially obviating the need for surgical interventions. However, it remains unclear whether topical application specifically exerts local or systemic effects in patients with axillary hyperhidrosis. This study's primary aim is to assess topical oxybutynin's impact on axillary hyperhidrosis.

Study Design: Twenty patients (initially planned sample size) diagnosed with axillary hyperhidrosis will be randomized into three groups. Group A will receive 2.5 mg of oral oxybutynin once daily at night for the first seven days, 2.5 mg twice daily from the 8th to the 21st day, and 5 mg twice daily from the 22nd to the 35th day. Group B will be administered a topical placebo as an oxybutynin spray, applying two sprays to each axilla twice daily for 35 days. Group C will receive a 10% oxybutynin topical spray, also used with two sprays to each axilla twice daily over 35 days (investigational product). The primary efficacy outcome will be the evaluation of the effectiveness of topical oxybutynin spray in treating hyperhidrosis, assessed by the number of patients showing an improvement in the severity of their condition by day 35, as measured by the Hyperhidrosis Disease Severity Scale (HDSS). Safety will be assessed by adverse and severe adverse events during the treatment

Summary: The TODAY trial will generate high-quality evidence on the effects of topical oxybutynin, assessing whether its impact is local or systemic in patients with axillary hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years and ≤ 45 years
* Not treated patient with another drug or treatment methodology for the disease for at least 30 days

Exclusion Criteria:

* Patients who are hypersensitive to oxybutynin hydrochloride.
* Not treated patient with another drug or treatment methodology for the disease for at least 30 days
* Patients who have menopausal symptoms
* Patients who show signs of skin lesions in the armpit
* Pregnancy. Women with the potential to bear children should be under contraceptive strategies and take a negative pregnancy test to be enrolled
* Patients with COVID in the contagious phase (PCR+)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in hyperhidrosis severity by day 35, as measured by the Hyperhidrosis Disease Severity Scale (HDSS) | Baseline and Day 35
  A treatment responder defined any participant whose HDSS score initially was 3 or 4 and who achieved at least a 1-point improvement in the scale by day 35.The HDSS is a patient completed validated scale that provides a qualitative measure of the severity of hyperhidrosis participants' condition based on how it affects their daily activities. It is a 4-point scale with scores defined as follows: 1 (underarm sweating was never noticeable and never interferes with daily activities); 2 (underarm sweating was tolerable but sometimes interferes with daily activities); 3 (underarm sweating was barely tolerable and frequently interferes with daily activities); and 4 (underarm sweating was intolerable and always interferes with daily activities). A score of 1 or 2 indicates mild or moderate hyperhidrosis. A score of 3 or 4 indicates severe hyperhidrosis.
Quality of life (QoL) assessment using the improvement metrics from a quality-of-life questionnaire published in 2003: de Campos JR et al. | From randomization to end of study at Day 35
  Mean improvement in QoL (Based on a 5 point scale with 0=no improvement and 5=extreme improvement). The difference between the final answer at the end of treatment at Day 35 and the one registered at baseline is called "the effect of treatment in the QOL".

SECONDARY OUTCOMES:
Clinical evaluation of adverse and severe adverse events was recorded as the number of participants experiencing adverse events, including dry mouth and cutaneous lesions. | Baseline and Day 35

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Ramacciotti, MD, PhD, Study Chair — Science Valley Research Institute
Locations (1):
- Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Red Cap open file.

REFERENCES:
- [Background] de Campos JR, Kauffman P, Werebe Ede C, Andrade Filho LO, Kusniek S, Wolosker N, Jatene FB. Quality of life, before and after thoracic sympathectomy: report on 378 operated patients. Ann Thorac Surg. 2003 Sep;76(3):886-91. doi: 10.1016/s0003-4975(03)00895-6. PMID 12963223
- [Background] Sharma P, Patel DP, Sanyal M, Berawala H, Guttikar S, Shrivastav PS. Simultaneous analysis of oxybutynin and its active metabolite N-desethyl oxybutynin in human plasma by stable isotope dilution LC-MS/MS to support a bioequivalence study. J Pharm Biomed Anal. 2013 Oct;84:244-55. doi: 10.1016/j.jpba.2013.06.024. Epub 2013 Jun 28. PMID 23867086